CLINICAL TRIAL: NCT03296891
Title: Randomized Point of Care Ultrasound Guided Resuscitation and Usual Care Comparison in the Management of Undifferentiated Shock: a Pilot Study
Brief Title: Point of Care Ultrasonography In The Management of Shock: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109038
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2017-09

CONDITIONS: Shock; Hypotension
Keywords: Ultrasonography; Point-of-care ultrasound; Resuscitation; Critical Care
MeSH Terms: conditions — Shock; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PoCUS Guided Resuscitation of Shock (Active Comparator): Participants randomized to this arm of the study will undergo PoCUS guided resuscitation of shock.
  Interventions: Other: PoCUS Guided Resuscitation of Shock
- Usual Care (No Intervention): Participants randomized to the 'usual care' arm of the study will be suggested to have the following guide resuscitation: 1) Pulse pressure variation (PPV), stroke volume variation (SVV) and/or systolic pressure variation (SPV) on their arterial line, 2) central venous pressure (CVP) and oxygen saturation(ScvO2) measurement, 3) Passive leg raise (PLR) maneuver, and/or 4) pulmonary artery catheter

INTERVENTIONS:
Other: PoCUS Guided Resuscitation of Shock — Point-of-care ultrasound (PoCUS) will be used to guide resuscitation of the participant with shock. A PoCUS study will consist of limited echocardiography (LE) and thoracic ultrasound (TUS).
  Arms: PoCUS Guided Resuscitation of Shock

SUMMARY:
This project aims to determine the feasibility of conducting a randomized controlled trial investigating point of care ultrasound guided resuscitation compared with usual care in the management of shock at the Critical Care Trauma Centre (CCTC) in London Health Science Centre (LHSC).

ELIGIBILITY:
Inclusion Criteria:

Patients deemed by the clinician to be in shock for any reason and has 3 out of 4 of the following:

1. Lactate greater than or equal to 2.2 mmol/L
2. AKIN stage I or greater or Urine output less than 0.5 cc/hr
3. Altered level of consciousness due to shock or requiring invasive mechanical ventilation as a result of shock
4. Vasoactive agents required to maintain a mean arterial pressure greater than 65 mmHg.

Exclusion Criteria:

1. Pregnant patients
2. Participants who have already undergone a PoCUS study (as defined in the protocol for this study) within the past 48 hours
3. Participants who have restrictions on their goals of care at the time of ICU admission (including patients refusing blood products).
4. Patients post cardiac arrest who are not obeying commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-07 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | averaged over 48 week period (active recruitment taking place in 48 of those 52 weeks)
  Number of patients who were successfully enrolled in the study per given week.

SECONDARY OUTCOMES:
Mortality | 28 days
  proportion of patients who are deceased for any reason at 28 days
Successful randomization rate | 28 days
  proportion of eligible patients who were randomized within the window for enrolment
Protocol adherence rate | 28 days
  Proportion of participants in the intervention arm that received the intended intervention
Contamination rate | 28 days
  Proportion of participants who were randomized to the control arm and inadvertently received the intervention
Revoked deferred consent rate | 28 days
  Proportion of participants whose consent was revoked
ICU length of stay | 28 days
  total days spent in ICU from time of admission to time of patient discharge
Ventilator free days | 28 days
  Days alive and free of mechanical ventilation at 28 days
Continuous renal replacement therapy free days | 28 days
  Days alive and free of vasoactive medications at 28 days
Vasoactive medication free days | 28 days
  Days alive and free of vasoactive medications at 28 days
Cumulative fluid balance | 7 days
  Fluid balance at 7 days post ICU admission or at time of discharge
Acute Kidney Injury (AKIN) stage | 7 days
  AKIN stage at 7 days post ICU admission or at time of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Science Center - Critical Care Trauma Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan for now to share individual participant data (IPD), but sharing anonymized data could be considered in the future.